CLINICAL TRIAL: NCT04289181
Title: A Pilot Trial Assessing the Feasibility of Providing Medically-tailored Meals to Patients Diagnosed With Heart Failure
Brief Title: A Trial to Evaluate Medically Tailored Meals With Patients With Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, AnnaMarie Chang, Associate Professor, Director of Clinical Research Operations, Thomas Jefferson University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 19G.837
Record Dates: First submitted 2020-02-17; First posted 2020-02-28 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Enrolled patients will be randomized to 1 of 2 arms: 1) MTM; or 2) usual care in a 1:1 ratio. A computer-generated list of random numbers will be prepared in advance by the study biostatistician and loaded into a REDCap randomization tool to ensure the research staff are blinded to assignment pre-randomization.
Masking Description: It is not feasible to blind participants and clinic staff to assignment post enrollment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medically Tailored Meals (MTM) (Experimental): Participants randomized to the MTM arm will receive MTM for 4 weeks. Meals will be prepared and delivered by Meals on Wheels, a non-profit organization that has been delivering meals to seniors nationwide for decades. Meals on Wheels will deliver 21 complete meals to the patient's home each week. They can accommodate a wide range of patient needs and preferences (e.g., low sodium, gluten-free, no pork products, cultural preferences). Meals on Wheels will contact the patient directly to set up an initial assessment phone call to collect relevant data (e.g., specific patient goals for their HF) and to set up a delivery schedule. Nearing the 4-week mark when meal delivery ends, investigators will check-in with each participant to track progress, assess treatment fidelity and answer any questions. All patients will receive information on community resources (e.g., food pantries, food banks) in the area.
  Interventions: Other: Medically Tailored Meals
- Usual Care (No Intervention): Patients in this arm will receive usual services offered at Jefferson for patients with HF. This includes regular visits with a HF provider (primary care or cardiology), standard nutrition teaching, medication optimization and post discharge support. During routine office visits, providers reinforce messages about self-management and provide lists of local and national resources related to nutrition and HF self-management. These services follow guideline directed medical therapy. All patients will receive information on community resources (e.g., food pantries, food banks) in the area.

INTERVENTIONS:
Other: Medically Tailored Meals — 4 weeks of medically tailored meals
  Arms: Medically Tailored Meals (MTM)

SUMMARY:
The goal is to conduct a pilot trial that provides 4 weeks of medically-tailored meals (MTM) to patients with heart failure (HF) via collaboration with the Philadelphia Meals on Wheels chapter to assess the feasibility of such an intervention. Patients will be enrolled during either an inpatient hospitalization or an emergency department (ED) visit, and will be randomized into 1 of 2 arms: 1) MTM or 2) usual care that follows guideline-directed medical therapy (GDMT). Evidence gathered from this study will guide the design of a larger randomized controlled trial to be submitted to the National Institutes of Health (NIH) to evaluate the scalability, sustainability and cost-effectiveness of MTM for improving outcomes for patients with HF.

DETAILED DESCRIPTION:
While medication adherence and transitions from hospitalization to home care play important roles in heart failure (HF) care, the majority of HF maintenance is by the patients in the home. Despite the availability of evidence-based guidance and treatments, many patients with HF do not achieve optimal outcomes. In prior work, patients with HF identified primary needs of improved access to food and nutrition education. Dietary recommendations for HF in clinical practice have historically emphasized the reduction of a single micronutrient (sodium) and fluid management, which oversimplifies the complexity between multiple dietary inadequacies, including micronutrient deficiencies, and HF pathophysiology. In addition, patients may have other comorbidities thus requiring further modification of the patient's diet. As a result, several innovative models for food services have emerged to address patient needs for improved healthy food access. Currently, select non-profit organizations across the U.S. deliver millions of medically-tailored meals (MTM) to patients with chronic illnesses, based on the premise that food can be as helpful as medicine in improving patient outcomes. Small studies assessing MTM in isolation have demonstrated reduced healthcare utilization and cost, however, no randomized trials have assessed the sustained impact of this intervention. The goal is to evaluate the feasibility of providing medically-tailored meals to patients with HF. Data from this study can be used to design further studies testing the effectiveness of MTM on improving outcomes for patients with HF.

Meals on Wheels, a provider of meals to senior citizens across the country, has only recently begun piloting medically-tailored meals, and this presents the opportunity to work with the organization to test the feasibility of MTM in the Philadelphia region.

ELIGIBILITY:
Inclusion Criteria:

1. Have a diagnosis of acute heart failure (AHF), as determined by the treating physician
2. Are 50 years of age or older
3. Are a patient in the ED or inpatient at TJUH or Methodist Hospita
4. Are able to keep food fresh for a week after delivery (e.g., not homeless)
5. Have an address that is within the delivery radius of Meals on Wheels-Philadelphia
6. Be able and willing to be available for follow-up contact

Exclusion Criteria:

1. Pregnant, planning to be pregnant, or currently breastfeeding.
2. Does not eat by mouth (i.e. receives tube feeds or total parenteral nutrition [TPN])
3. Psychiatric co-morbidity that would preclude study participation
4. Non-English speaking
5. In police custody or incarcerated
6. Currently receiving MTM from Meals on Wheels or another provider

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Feasibility: Enrollment | One year
  Feasibility will be measured by the number of patients enrolled in the study. We aim to enroll 30 total patients.
Feasibility: Retention | 4 weeks
  Feasibility will be measured by the percent of enrolled patients who complete follow-up visits at 4 weeks
Feasibility: Retention | 12 weeks
  Feasibility will be measured by the percent of enrolled patients who complete follow-up visits at 12 weeks

SECONDARY OUTCOMES:
Patient satisfaction with intervention | 4 weeks
  Satisfaction will be measured using a series of satisfaction related questions to better understand patients' experience with receiving medically tailored meals. Likert scale questions will be asked upon the completion of the meal deliveries at the 4 week follow-up assessment. Questions will assess the convenience, taste, and size of received meals.
Feasibility of administering the patient activation measure short form (PAM-13) | Baseline, 4 weeks, 12 weeks
  The PAM-13 is composed of 13 items measuring patients' self-reported knowledge, motivation, and skills for health management. Each item is measured on a 5-point likert scale from disagree strongly to agree strongly. Those who score lower on the scale have lower self-management skills, while those who score higher on the scale are more engaged in their self-management.
Feasibility of administering the Dutch Heart Failure Knowledge Scale | Baseline, 4 weeks, 12 weeks
  The Dutch Heart Failure Knowledge Scale consists of 15 multiple choice questions assessing knowledge about Heart Failure in general (4 items), treatment (6 items), and symptoms and symptom recognition (5 items). Patients are instructed to choose the correct response from the three choices provided. The assessment is scored from 0 (no knowledge) to 15 (optimal knowledge).
Feasibility of administering the Kansas City Cardiomyopathy Questionnaire 12 (KCCQ-12) | Baseline, 4 weeks, 12 weeks
  The KCCQ-12, a self-administered 12-item instrument, assesses physical limitations, symptoms, self-efficacy, social interference, and overall quality of life (QoL) in HF patients. Higher scores on the KCCQ-12 indicate better QoL. The KCCQ summary score independently predicts clinical outcomes such as hospitalization and mortality in outpatients with HF, including those recently hospitalized for acute decompensation. It is a reliable and valid measure in HF patients that is more sensitive to change than other measures of QoL, and is especially responsive in patients with multiple comorbidities. A change in KCCQ score of 5 points is clinically significant and correlates with changes in clinical status, physical function, and outcomes.
Feasibility of administering the Minnesota Living with Heart Failure Questionnaire (MLHF) | Baseline, 4 weeks, 12 weeks
  The MLHF measures the effects of heart failure and treatments for heart failure on an individual's quality of life. The questionnaire includes 21 items scored on a 6-point likert scale from zero (no impact) to five (big impact). All questions ask the patient to identify how much HF has affected their life during the past month. The survey is scored by adding all 21 responses for a total score. A physical dimension score (8 items) and emotional dimension score (5 items) can also be derived by adding the scores for specific items.

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States